CLINICAL TRIAL: NCT04049890
Title: Development and Validation of a New Instrument to Evaluate Parents' Adjustment to Their Child's Chronic Disease: the Family Adjustment Inventory
Brief Title: Development and Validation of Family Adjustment Inventory
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Pediatric Psychologist, Meyer Children's Hospital IRCCS
Other Study IDs: FAI
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-10

CONDITIONS: Adjustment Reaction
Keywords: adjustment; family functioning; chronic disease; emotions
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parents of children with a chronic disease with no siblings: Parents of children suffering from a chronic disease who has no brother or sister over 3 years of age
  Interventions: Other: FAI-O; Other: Personal Data Questionnaire
- Parents of children with a chronic disease with siblings: Parents of children suffering from a chronic disease who one or more sibling over the age of 3 years old
  Interventions: Other: FAI-S; Other: Personal Data Questionnaire

INTERVENTIONS:
Other: FAI-O — Administration of Family Adjustment Inventory in the version "Only-child"
  Groups: Parents of children with a chronic disease with no siblings
Other: FAI-S — Administration of Family Adjustment Inventory in the version "Sibling"
  Groups: Parents of children with a chronic disease with siblings
Other: Personal Data Questionnaire — This form requires informations about child, respondent and partner (if any), and evaluates the presence of any distressful event happened during the last year

SUMMARY:
A diagnosis of chronic disease in childhood may be disruptive for families. Some parents show good adjustment, while others may have more difficulties.

Aim of this study is to develop and validate a new psychometric instrument to help precociously detect parents' vulnerability in the process of adjustment to their child's chronic disease at different times of care.

DETAILED DESCRIPTION:
FAI was developed in two different forms:

1. for parents with one children suffering from a chronic disease or ill children who has siblings younger than 3 years old - FAI-O (only child);
2. for parents with at least two children, the brother/sister of the ill child has 3 years or more- FAS-S (siblings) The two forms are identical, with the exception that FAI-S has an additional dimension with respect to FAI-O, that specifically regards the involvement of siblings in the illness path of the sick brother/sister.

Development of FAI followed several steps:

* definition of initial instrument dimensions
* item wording for each dimension
* definition of scoring
* focus group with parents of patients suffering from a chronic disease to evaluate item content and linguistic clarity

Validation of FAI for each form (FAI-O and FAI-S):

Validation consists in several steps, identical for the two versions but in different in timing, depending on the number of admnistration.

* first phase: the FAI is administered to parents of patients with different chronic disease (each form needs to reach the total of 300 administrations).
* second phase: statistical analysis aimed to obtain the final version of each FAI form (define actual dimensions and most adequate items)
* third phase: administration to a new sample of parents of children suffering from a chronic disease (each form needs to reach the total of 150 administrations).
* fourth phase: statistical analysis aimed to confirm the adequacy of the instrument

ELIGIBILITY:
Inclusion Criteria:

* consent for participating in the study
* having a child suffering from a chronic illness and treated in the hospital in the following specialties: onco-hematology, neuro-oncology, diabetology, cystic fibrosis, metabolic disease, gastroenterology, cardiology, nephrology, rheumatology, allergology, pneumology, immunology, intensive care unit
* italian speaking

Exclusion Criteria:

* cognitive impairment
* no good knowledge of italian language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of patient with a child sufferinf from a chronic illness and treated in the hospital for this condition .
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-03-15 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Perceived family adjustment | Parents fill in the FAI one single time at enrollment
  FAI (Family Adjustment Inventory) measures family adjustment. The preliminary versions of FAI-O consists in182 items and FAI-S in197 items, both scored on a 5-point likert scale from 0 to 4. Higher scores represent poorer adjustment.

SECONDARY OUTCOMES:
Presence of distressful events happened in the last year | Parents fill in the personal data questionnaire one single time at enrollment
  The presence of distressful events is collected through a personal data questionnaire, specifically designed for this study in accordance to literature in the field

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Maffei, Msc, Study Director — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children's Hospital, Florence, Firenze, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aneshensel CS, Pearlin LI, Mullan JT, Zarit SH, Whitlatch CJ (1995). Profiles in caregiving: the unexpected career. San Diego Academic Press, Inc.
- [Background] Boer LM, Daudey L, Peters JB, Molema J, Prins JB, Vercoulen JH. Assessing the stages of the grieving process in chronic obstructive pulmonary disease (COPD): validation of the Acceptance of Disease and Impairments Questionnaire (ADIQ). Int J Behav Med. 2014 Jun;21(3):561-70. doi: 10.1007/s12529-013-9312-3. PMID 23645551
- [Background] Bonner MJ, Hardy KK, Guill AB, McLaughlin C, Schweitzer H, Carter K. Development and validation of the parent experience of child illness. J Pediatr Psychol. 2006 Apr;31(3):310-21. doi: 10.1093/jpepsy/jsj034. Epub 2005 May 25. PMID 15917492
- [Background] Klassen AF, Raina P, McIntosh C, Sung L, Klaassen RJ, O'Donnell M, Yanofsky R, Dix D. Parents of children with cancer: which factors explain differences in health-related quality of life. Int J Cancer. 2011 Sep 1;129(5):1190-8. doi: 10.1002/ijc.25737. Epub 2010 Dec 17. PMID 21064097
- [Background] McCubbin HI, McCubbin MA, Patterson JM, Cauble AE, Wilson LR, Warwick W. (1983). CHIP Coping Health Inventory for Parents: an assessment of parental coping patterns in the care of the chronically ill child. Journal of Marriage and Family, 45(2), 359-370.
- [Background] Raina P, O'Donnell M, Schwellnus H, Rosenbaum P, King G, Brehaut J, Russell D, Swinton M, King S, Wong M, Walter SD, Wood E. Caregiving process and caregiver burden: conceptual models to guide research and practice. BMC Pediatr. 2004 Jan 14;4:1. doi: 10.1186/1471-2431-4-1. PMID 14723791
- [Background] Raina P, O'Donnell M, Rosenbaum P, Brehaut J, Walter SD, Russell D, Swinton M, Zhu B, Wood E. The health and well-being of caregivers of children with cerebral palsy. Pediatrics. 2005 Jun;115(6):e626-36. doi: 10.1542/peds.2004-1689. PMID 15930188
- [Background] Rossi Ferrario S, Baiardi P, Zotti AM. Update on the family strain questionnaire: a tool for the general screening of caregiving-related problems. Qual Life Res. 2004 Oct;13(8):1425-34. doi: 10.1023/B:QURE.0000040795.78742.72. PMID 15503838